CLINICAL TRIAL: NCT04567225
Title: Early Basal Insulin Administration in Adult Diabetic Ketoacidosis Management
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped after internal review
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Mohammed Al-Jaghbeer, Clinical Assistant professor and Principal Investigator, The Cleveland Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-903
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Results first posted 2022-08-25 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Ketoacidosis; Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetic Ketoacidosis; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Fluid Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Early Glargine (Experimental): All consecutive adult patients getting admitted to Medical ICU and meet the inclusion criteria and accepted to receive insulin glargine early as per the protocol. They will receive insulin glargine 0.4 unit/kg within 4 hours from initiating the IV Insulin Infusion, as per the Cleveland Clinic DKA protocol.
  Interventions: Drug: Early Glargine; Other: IV insulin infusion; Other: IV fluid and electrolytes replacement
- Standard practice (Late Glargine) (Active Comparator): Retrospective, prespecified and matched sample of consecutive adults who admitted to the same Medical ICU with a diagnosis of DKA in the period between January 1st 2019 till the Institutional Review Board (IRB) approval date and didn't receive basal insulin before Anion Gap closure.
  Interventions: Drug: Late Glargine; Other: IV insulin infusion; Other: IV fluid and electrolytes replacement

INTERVENTIONS:
Drug: Early Glargine — A dose of insulin glargine, 0.4 unit/kg, will be given within 4 hours from initiating the IV Insulin Infusion
  Other Names: lantus
  Arms: Early Glargine
Drug: Late Glargine — A historical retrospective control group for the adult patients admitted to the same ICU with a diagnosis of DKA and received insulin glargine after anion gap closure.
  Other Names: lantus
  Arms: Standard practice (Late Glargine)
Other: IV insulin infusion — Continuous weight based IV insulin infusion as per Cleveland Clinic DKA Protocol
Other: IV fluid and electrolytes replacement — The IV fluid and electrolytes replacement will be left to the treating physician's discretion. IV fluid to contain dextrose to keep Target Blood Glucose 150 - 200 mg/dl during the DKA management and 140 - 180 mg/dl after DKA resolution.

SUMMARY:
Early Basal Insulin Administration in Adult Diabetic Ketoacidosis Management

DETAILED DESCRIPTION:
The transition from IV Insulin Infusion (IVII) to Subcutaneous Long-acting insulin injections in Diabetic Ketoacidosis (DKA) management frequently results in rebound hyperglycemia, particularly if there are high insulin requirements that can adversely affect the DKA recovery, increase Length Of Stay (LOS), morbidity, and mortality. Investigators propose a prospective, open-label, intervention, non-randomized, controlled study to test the hypothesis that an insulin glargine dose of 0.4 Units/kg early administered (within four hours) of IVII initiation in DKA management in adult would be effective and safe in shortening the time to anion gap closure comparing to the standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Meet DKA definition (BG ≥ 250 mg/dl, Anion Gap > 12 mEq/L, and positive Ketones in serum or urine)
* Having the capacity to sign Informed consent

Exclusion Criteria:

* IV insulin infusion was initiated for more than 4 hours.
* Persistent hypotension (SBP<80 mmHg despite receiving 1000cc normal saline).
* Require Vasopressor
* Acute Coronary Syndrome
* Pregnant
* End-stage renal disease
* Unwilling to consent to participate in the trial
* Currently under police custody
* Transferred from another hospital
* Require emergent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Al jaghbeer, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Fairview Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Individual subject results will not be shared with those involved in the prospective arm

REFERENCES:
- [Background] Realsen J, Goettle H, Chase HP. Morbidity and mortality of diabetic ketoacidosis with and without insulin pump care. Diabetes Technol Ther. 2012 Dec;14(12):1149-54. doi: 10.1089/dia.2012.0161. Epub 2012 Sep 25. PMID 23009106
- [Background] Kitabchi AE, Umpierrez GE, Miles JM, Fisher JN. Hyperglycemic crises in adult patients with diabetes. Diabetes Care. 2009 Jul;32(7):1335-43. doi: 10.2337/dc09-9032. No abstract available. PMID 19564476
- [Background] Bunn S, Halm M. Long-Acting Insulin on the Road to Recovery With Diabetic Ketoacidosis. Am J Crit Care. 2016 May;25(3):277-80. doi: 10.4037/ajcc2016681. No abstract available. PMID 27134235
- [Background] Hsia E, Seggelke S, Gibbs J, Hawkins RM, Cohlmia E, Rasouli N, Wang C, Kam I, Draznin B. Subcutaneous administration of glargine to diabetic patients receiving insulin infusion prevents rebound hyperglycemia. J Clin Endocrinol Metab. 2012 Sep;97(9):3132-7. doi: 10.1210/jc.2012-1244. Epub 2012 Jun 8. PMID 22685233
- [Background] Savage MW, Dhatariya KK, Kilvert A, Rayman G, Rees JA, Courtney CH, Hilton L, Dyer PH, Hamersley MS; Joint British Diabetes Societies. Joint British Diabetes Societies guideline for the management of diabetic ketoacidosis. Diabet Med. 2011 May;28(5):508-15. doi: 10.1111/j.1464-5491.2011.03246.x. PMID 21255074
- [Background] Doshi P, Potter AJ, De Los Santos D, Banuelos R, Darger BF, Chathampally Y. Prospective randomized trial of insulin glargine in acute management of diabetic ketoacidosis in the emergency department: a pilot study. Acad Emerg Med. 2015 Jun;22(6):657-62. doi: 10.1111/acem.12673. Epub 2015 May 25. PMID 26013711
- [Background] Houshyar J, Bahrami A, Aliasgarzadeh A. Effectiveness of Insulin Glargine on Recovery of Patients with Diabetic Ketoacidosis: A Randomized Controlled Trial. J Clin Diagn Res. 2015 May;9(5):OC01-5. doi: 10.7860/JCDR/2015/12005.5883. Epub 2015 May 1. PMID 26155506
- [Background] Shankar V, Haque A, Churchwell KB, Russell W. Insulin glargine supplementation during early management phase of diabetic ketoacidosis in children. Intensive Care Med. 2007 Jul;33(7):1173-1178. doi: 10.1007/s00134-007-0674-3. Epub 2007 May 17. PMID 17508198

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was closed due to lack of proper resource availability. Since study could not be completed as planned, no analysis was completed. This included no enrollment into the chart review arm.
Groups:
- Early Glargine: All consecutive adult patients getting admitted to Medical ICU and meet the inclusion criteria and accepted to receive insulin glargine early as per the protocol. They will receive insulin glargine 0.4 unit/kg within 4 hours from initiating the IV Insulin Infusion, as per the Cleveland Clinic DKA protocol.
  Glargine: A dose of insulin glargine, 0.4 unit/kg, will be given within 4 hours from initiating the IV Insulin Infusion
  IV insulin infusion: Continuous weight based IV insulin infusion as per Cleveland Clinic DKA Protocol
  IV fluid and electrolytes replacement: The IV fluid and electrolytes replacement will be left to the treating physician's discretion. IV fluid to contain dextrose to keep Target Blood Glucose 150 - 200 mg/dl during the DKA management and 140 - 180 mg/dl after DKA resolution.
- Standard Practice (Late Glargine): Retrospective, prespecified and matched sample of consecutive adults who admitted to the same Medical ICU with a diagnosis of DKA in the period between January 1st 2019 till the Institutional Review Board (IRB) approval date and didn't receive basal insulin before Anion Gap closure.
  Glargine: A historical retrospective control group for the adult patients admitted to the same ICU with a diagnosis of DKA and received insulin glargine after anion gap closure.
  IV insulin infusion: Continuous weight based IV insulin infusion as per Cleveland Clinic DKA Protocol
  IV fluid and electrolytes replacement: The IV fluid and electrolytes replacement will be left to the treating physician's discretion. IV fluid to contain dextrose to keep Target Blood Glucose 150 - 200 mg/dl during the DKA management and 140 - 180 mg/dl after DKA resolution.
Period: Overall Study
Arm/Group | Early Glargine | Standard Practice (Late Glargine)
Started | 39 | 0
Completed | 0 (Study withdrawn. The study was closed due to lack of proper resource availability. Since study could not be completed as planned, participants did not complete follow-up.) | 0 (The study was closed due to lack of proper resource availability. Since study could not be completed as planned, this chart review portion was not completed and no analysis was performed.)
Not Completed | 39 | 0

BASELINE CHARACTERISTICS:
Population: Study withdrawn. The study was closed due to lack of proper resource availability. Since study could not be completed as planned, no analysis was completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Glargine | Standard Practice (Late Glargine) | Total
Number analyzed (Participants) | 39 | 0 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 0 | 31
  >=65 years | 8 | 0 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 0 | 20
  Male | 19 | 0 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 0 | 10
  Not Hispanic or Latino | 29 | 0 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 11 |  | 11
  White | 21 |  | 21
  More than one race | 0 |  | 0
  Unknown or Not Reported | 7 |  | 7
Region of Enrollment [Number; unit: participants]
  United States | 39 |  | 39

OUTCOME MEASURES:

1. Primary Outcome: Time to Anion Gap Closure
Description: Measured in hours from starting insulin infusion till anion gap ≤ 12 milliequivalent/Liter (mEq/L)
Time Frame: Participants monitored from hospital admission to discharge, an average of 5 days
Population: Study withdrawn. The study was closed due to lack of proper resource availability. Since study could not be completed as planned, no data was collected for analysis.
Arm/Group | Early Glargine | Standard Practice (Late Glargine)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Hospital Length of Stay
Description: The time, in days, from the patient admission to the hospital till discharge
Time Frame: Participants monitored from hospital admission to discharge, an average of 5 days
Population: as for outcome 1
Arm/Group | Early Glargine | Standard Practice (Late Glargine)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: ICU Length of Stay
Description: The time, in hours, from the patient admission to the ICU till transfer to regular nursing floor
Time Frame: Participants monitored from hospital admission to discharge, an average of 5 days
Population: as for outcome 1
Arm/Group | Early Glargine | Standard Practice (Late Glargine)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Total IV Insulin Infusion Dose
Description: the total amount of insulin infusion, by International Unit, has been received by the patient during the DKA treatment
Time Frame: Participants monitored from hospital admission to discharge, an average of 5 days
Population: as for outcome 1
Arm/Group | Early Glargine | Standard Practice (Late Glargine)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Incidence of Transitional Failure
Description: Defined as the recurrence of DKA (BG ≥ 250 mg/dl, Anion Gap > 12 milliequivalent/Liter (mEq/L), and positive Ketones in serum or urine) after initial IV insulin infusion (IVII) discontinuation within 24 hours and requiring re-initiating the IVII
Time Frame: up to 24 hours after IVII discontinuation
Population: as for outcome 1
Arm/Group | Early Glargine | Standard Practice (Late Glargine)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Incidence of Hyperglycemia
Description: Incidence of hyperglycemia (> 180 mg/dL) after IVII discontinuation
Time Frame: up to 24 hours after initial Insulin Glargine dose
Population: as for outcome 1
Arm/Group | Early Glargine | Standard Practice (Late Glargine)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Incidence of Hypoglycemia
Description: Incidence of hypoglycemia (defined as ≤ 70 mg/dL, <54 mg/dL, <40 mg/dl) after IVII discontinuation
Time Frame: up to 24 hours after initial Insulin Glargine dose
Population: as for outcome 1
Arm/Group | Early Glargine | Standard Practice (Late Glargine)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Consent through date of discharge (an average of 5 days)
Description: No patients were enrolled in the Standard Practice (Late Glargine) arm.
Arm/Group | Early Glargine | Standard Practice (Late Glargine)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/0
Other Adverse Events (participants affected / at risk) | 0/39 | 0/0

LIMITATIONS AND CAVEATS:
The study was closed due to lack of proper resource availability. Since study could not be completed as planned, no analysis was completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT04567225/Prot_SAP_000.pdf